CLINICAL TRIAL: NCT06672081
Title: A Randomized Trial for Early Catheter-directed Treatment of High Risk Pulmonary Embolism
Brief Title: Early Catheter-directed Treatment of High Risk Pulmonary Embolism
Acronym: CATCH-PE II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leipzig Heart Science gGmbH (Other)
Collaborators: Heart Center Leipzig at University of Leipzig (Unknown); Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0124
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Embolism Acute Massive
Keywords: pulmonary embolism; early catheter-directed treatment
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional care (Active Comparator): Patients in the conventional care group will receive guideline directed therapy including reperfusion treatment. If no clinically relevant hemodynamic improvement occurs, catheter-interventional treatment may be used as stated in the current ESC-guidelines
  Interventions: Drug: Conventional care
- Early Catheter-Interventional Treatment + conventional care (Experimental): Patients in this group will undergo a catheter-interventional treatment within 60 min. after randomization. Fibrinolytic treatment will be prepared parallel to interventional treatment preparations to avoid any delay in its administration, if clinically necessary. Catheter-interventional treatment may include any certified devices for the treatment of PE including aspiration thrombectomy, local fibrinolytic therapy, local ultrasound treatment as assistance to local fibrinolysis or any combination of these. Transfemoral venous access routes will be used for any catheter-directed treatment using sheath-sizes as recommended in the IFUs by the respective manufacturers. Sheaths will be withdrawn immediately after catheter-based thrombectomy or after completion of catheter-directed local fibrinolysis, typically 5 to 10 hours after initiation. The choice of the catheter types and sizes will be left to the treating interventionalists' discretion.
  Interventions: Procedure: Early Catheter-Interventional Treatment; Drug: Conventional care

INTERVENTIONS:
Procedure: Early Catheter-Interventional Treatment — Patients will undergo a catheter-interventional treatment within 60 min. after randomization. Fibrinolytic treatment will be prepared parallel to interventional treatment preparations to avoid any delay in its administration if clinically necessary. Catheter-interventional treatment may include any certified devices for the treatment of PE including aspiration thrombectomy, local fibrinolytic therapy, local ultrasound treatment as assistance to local fibrinolysis or any combination of these.Transfemoral venous access routes will be used for any catheter-directed treatment using sheath-sizes as recommended in the IFUs by the respective manufacturers. Sheaths will be withdrawn immediately after catheter-based thrombectomy or after completion of catheter-directed local fibrinolysis, typically 5 to 10 hours after initiation.
  Arms: Early Catheter-Interventional Treatment + conventional care
Drug: Conventional care — reperfusion treatment

SUMMARY:
Prospective, multicenter, open label, randomized controlled clinical trial to compare the effects of an early catheter-directed treatment plus conventional care with conventional care in patients with high-risk pulmonary embolism

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary embolism as confirmed by CT angiogram with high mortality risk as defined by ESC guidelines:

   a) One of the following: i. Cardiac arrest or ii. obstructive shock (systolic BP <90 mmHg or vasopressors required to achieve a BP ≥90 mmHg despite an adequate filling status), in combination with end-organ hypoperfusion (cold, clammy skin, oliguria or serum lactate ≥2 mmol/L) and b) Signs of right-ventricular dysfunction on transthoracic echocardiogram or CT scan
2. Age ≥18 years

Exclusion Criteria:

1. Contraindications for catheter-based treatment
2. Contraindications to systemic fibrinolytic treatment or anticoagulation*

   1. Active, potentially life-threatening bleeding
   2. Surgery within 24h before screening
   3. Cranial or spinal surgery within 14d before screening
   4. Stroke within 14d before screening
   5. Intracranial tumor
   6. Any condition not listed here but estimated as clinically relevant as judged by the treating investigator
3. Pregnancy

   * Patients with contraindications to systemic fibrinolysis or anticoagulation can be enrolled in a third study arm (registry) and undergo catheter-directed therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of mortality (all-cause) and recurrent cardiac arrest or persistent / recurrent shock | 7 days
  1. mortality (all-cause) up to 7 days after randomization and
  2. either one of the following
     1. recurrent cardiac arrest or
     2. persistent / recurrent shock (systolic BP <90 mmHg or vasopressors or ECMO required to achieve a systolic BP ≥90 mmHg, in combination with end-organ hypoperfusion (cold, clammy skin, oliguria or serum lactate ≥2 mmol/L) 24 hours after randomization

SECONDARY OUTCOMES:
All-cause mortality | 7 days
  All-cause mortality at day 7 after randomization
PE-related mortality | 7 days
  PE-related mortality at day 7 after randomization
Mortality (all-cause) | 30 days
  Mortality (all-cause) at day 30 after randomization
Bail out therapy | 7 days
  Bail out therapy at day 7 after randomization
GUSTO moderate or severe bleeding | 7 days
  GUSTO moderate or severe bleeding up to 7 days after randomization
VA-ECMO use | 7 days
  VA-ECMO use between randomization and day 7 after randomization
Change in echocardiographic parameters | 24 hours
  Change in echocardiographic parameters (RV/LV ratio, RV-strain, TAPSE) 24h after randomization
Days of ICU stay | 30 days
  Days of ICU stay
Time to hemodynamic stabilization | 30 days
  Time to hemodynamic stabilization

CONTACTS AND LOCATIONS:
Overall Officials: Karl Fengler, MD, Assoc. Prof., Study Chair — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology; Holger Thiele, MD. Prof., Study Chair — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology
Locations (11):
- Germany (11):
  - Universitätsklinikum Freiburg, Bad Krozingen
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Halle, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - SLK-Kliniken Heilbronn, Heilbronn
  - Universitätsklinikum Leipzig, Leipzig
  - Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology, Leipzig
  - Universitätsklinikum Mannheim, Mannheim
  - Schwarzwald-Baar-Klinikum, Villingen-Schwenningen
  - Rems-Murr-Kliniken, Winnenden
  - Helios Kliniken Wuppertal, Wuppertal

IPD SHARING:
Plan to Share IPD: No